CLINICAL TRIAL: NCT01357434
Title: Rating Fast Food on Healthiness
Brief Title: Comparing Calories at Fast Food Restaurants
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Lenard I Lesser, University of California, Los Angeles
Other Study IDs: RAND2010-0808
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents: Participants 12-21 years old.
  Interventions: Behavioral: Fast Food Restaurant

INTERVENTIONS:
Behavioral: Fast Food Restaurant — Participants will purchase a meal at Subway and McDonald's, on different days.

SUMMARY:
Rating systems are intended to guide consumer choices. This project will determine if a previously developed scale that evaluates the "healthiness" of a restaurant is correlated with the actual choices consumers make when they patronize the restaurants. The study will also assess whether a restaurant marketed as "healthy" (Subway) rates higher on this scale than another restaurant that makes no such claims (McDonald's). Finally, the investigators will compare the calorie purchases from these two restaurants among youths and their families who eat at each of the restaurants.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 Year Olds that live in local area
* Like to eat at Subway and McDonald's

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents in a community in South Los Angeles.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Calories Consumed at each Restaurant | Calories will be recorded at two time points within 1-2 weeks
  Using purchase receipts and point-of-purchase surveys, we determine how many calories each participant purchases.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, University of California, Los Angeles, California, United States

REFERENCES:
- [Derived] Lesser LI, Kayekjian KC, Velasquez P, Tseng CH, Brook RH, Cohen DA. Adolescent Purchasing Behavior at McDonald's and Subway. J Adolesc Health. 2013 Oct;53(4):441-5. doi: 10.1016/j.jadohealth.2013.02.014. Epub 2013 May 6. PMID 23660412